## POWER ANALYSIS REPORT

Statistical power analysis was applied to decide how many observations to work with for the article study on "An Evaluation of the Effect of Grain-Like Products on Postprandial Glucose, Insulin and Subjective Saturation Response in Healthy Individuals". For power analysis, power values for different sample numbers were calculated with G\*Power software. While calculating the power values, the results were determined within the scope of 95% confidence level (p<0.05). Parallel to the research to be carried out, starting from the reference study (Vuksan et al., 2017), the independent samples t-test result applied to describe the mean difference in waist circumference was taken as a basis. The effect size value obtained for the power analysis within the scope of the applied test was calculated as approximately d=3.429. According to the power values, in this study, if a total of 6 observations are studied, a test power of approximately 87.4% is reached. Since the power value we calculated is over 80%, it is statistically sufficient. Figure 1 shows the graph of power values according to the number of samples. In addition, the screen output of the G\*Power program is given in Figure 2.



Figure 1: Power values for different sample numbers

```
Post hoc: Compute achieved power
Analysis:
Input:
             Tail(s)
                                                     Two
                                                     3.428571
             Effect size d
             α err prob
                                                     0.05
             Sample size group 1
             Sample size group 2
                                                     3
Output:
             Noncentrality parameter \delta
                                                     4.1991247
             Critical t
                                                     2.7764451
             Df
             Power (1-\beta \text{ err prob})
                                                     0.8741037
```

**Figure 2:** G\*Power screen output

## Reference

Vuksan V, Jenkins AL, Brissette C, Choleva L, Jovanovski E, Gibbs AL, Bazinet RP, Au-Yeung F, Zurbau A, Ho HV, Duvnjak L, Sievenpiper JL, Josse RG, Hanna A. Salba-chia (Salvia hispanica L.) in the treatment of overweight and obese patients with type 2 diabetes: A double-blind randomized controlled trial. Nutr Metab Cardiovasc Dis. 2017 Feb;27(2):138-146. doi: 10.1016/j.numecd.2016.11.124. Epub 2016 Dec 9. PMID: 28089080.